CLINICAL TRIAL: NCT06848465
Title: A Phase Ib Trial on the Safety and Feasibility of Low Dose Radiotherapy (LDRT) Combined With Immunochemotherapy for Colorectal Cancer With Liver-limited Metastasis
Brief Title: LDRT Combined With Immunochemotherapy for Colorectal Cancer With Liver Metastasis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DP2024348
Record Dates: First submitted 2025-01-22; First posted 2025-02-27 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-02

CONDITIONS: Colorectal Cancer; Liver Metastasis; LDRT
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Radiotherapy; XELOX; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LDRT/LDRT+SCRT followed by Tislelizumab+XELOX (Experimental): For patients with colon Cancer:
  LDRT starts from day 1.
  For patients with rectal Cancer:
  LDRT and SCRT start concurrently from day 1. Tislelizumab+XELOX start from 1week after the completion of radiotherapy (2-4 cycles).
  Interventions: Radiation: Low Dose Radiotherapy; Radiation: Short course Radiotherapy; Drug: XELOX; Drug: Tislelizumab

INTERVENTIONS:
Radiation: Low Dose Radiotherapy — 10 Gy in 5 fractions, 15 Gy in 3 fractions, 20 Gy in 10 fractions respectively in three Cohorts from Day1
Radiation: Short course Radiotherapy — 25 Gy in 5 fractions from Day1
Drug: XELOX — Oxaliplatin: 130mg/m2 IV Q3W on day 1 of each cycle. Capecitabine: 1000mg/m2 Q3W Dose of 1000mg/m2 on day 1-14 of each cycle.
Drug: Tislelizumab — 200mg IV Q3W on day 1 of each cycle.

SUMMARY:
In recent years, growing evidences have demonstrated promising synergistic antitumor effects of radiotherapy combined with immunotherapy. More over, LDRT may enhance the antitumor effect of immunotherapy by altering the tumor immune microenvironment (TIME) and adjusting the immune response. In this study, we will explore the safety and feasibility of LDRT and immunochemotherapy in liver metastatic colorectal cancer. 9-18 participants will be enrolled in this study. All will take part at Daping Hospital, Army Medical University.

DETAILED DESCRIPTION:
This is a prospective, single-arm, phase Ib trial. At least 9 eligible patients will be will be enrolled In this study. Patients will receive LDRT of 10 Gy in 5 fractions, 15 Gy in 5 fractions, 20 Gy in 10 fractions respectively in our three groups on liver metastsis from Day1 (patients with rectal cancer will receive SCRT concurrently), followed by Xelox and Tislelizumab starting from 1 week after the completion of radiation. The primary endpoints are safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

1. Age between18 and 75 years old.
2. Histopathological confirmed MSS/pMMR adenocarcinoma of the colon or rectum.
3. The clinical baseline stage of rectal cancer assessed by MRI/CT/Transrectal ultrasound was T3-4Nx or TXN1-2.
4. Simultaneous liver metastasis confirmed by imaging examination.
5. No previous antitumor treatment.
6. An Eastern Cooperative Oncology Group (ECOG) performance status ≤1.
7. Adequate cardiac function (Left Ventricular Ejection Fractions > 50%), hepatic function (total serum bilirubin ≤ 1.5 × upper limit of normal, alanine aminotransferase or aspartate aminotransferase ≤ 2.5 × upper limit of normal), renal function (serum creatinine ≤ 1.5 × ULN or glomerular filtration rate > 60 ml/min, based on Cockcroft-Gault), and hematopoietic function (white blood cells ≥ 4.0 × 109 cells per L, neutrophils ≥ 1.5 × 109 cells per L, hemoglobin ≥ 90 g/L, platelets ≥ 100 × 109 cells per L).
8. Sign the informed consent and have good compliance.

Exclusion Criteria:

1. Distant metastasis from other than the liver.
2. BMI < 18.5 kg/m² or weight loss ≥ 10% within the past 6 months (with consideration of the impact of large amounts of pleural and ascitic fluid on body weight).
3. Received any of the following treatments: any investigational drug; enrolled in another clinical trial concurrently, unless it is an observational (non-interventional) clinical study; received anti-tumor vaccines or live vaccines.
4. Active autoimmune diseases, or a history of autoimmune diseases. A history of liver disease including, but not limited to HBV infection or HBV DNA positive(≥1×10^4/ml), HCV infection or HCV DNA positive(≥1×10^3/ml) and liver cirrhosis.
5. History of immunodeficiency, including positive HIV test, or other acquired or congenital immunodeficiency diseases, or history of organ transplantation and allogeneic bone marrow transplantation.
6. A history of heart disease within 6 months (including congestive heart failure, acute myocardial infarction, severe/unstable angina, coronary artery bypass grafting, cardiac insufficiency ≥ NYHA grade 2 and LVEF<50%).
7. The presence of a clinically detectable second primary malignancy, or history of other malignancies within 5 years excluding adequately treated non-melanoma skin cancer, carcinoma in situ of cervix and superficial bladder tumour (non-invasive tumour, or carcinoma in situ, or T1).
8. Pregnant or lactating women.
9. The investigator considers that the subject is not suitable to participate in this clinical study due to any clinical or laboratory abnormalities or compliance problems.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | 3 years
  Number of participants with Adverse Events and/or Dose Limiting Toxicities as a Measurement of Safety and tolerability of LDRT in Combination With Tirellizumab and XELOX

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 2 years
  Investigator assessed ORR using RECIST v1.1 including the all tumor
Progression-free survival (PFS) | 2 years
  Defined as the time from initiation of treatment to tumor progression or death from any cause.
Overall survival (OS) | 3 years
  Defined as the time from initiation of treatment to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Chuan Chen, MD PhD, Study Director — Daping Hospital, Army Medical University
Locations (2):
- China (2):
  - Army Medical Center, Chongqing, Chongqing Municipality
  - Daping Hospital, Army Medical University, Chongqing, Chongqing Municipality

IPD SHARING:
Plan to Share IPD: No